CLINICAL TRIAL: NCT02211053
Title: Evaluation of the Efficacy and Safety of Levothyroxine in Brain Death Organ Donors: a Randomized Controlled Trial
Brief Title: Evaluation of the Efficacy and Safety of Levothyroxine in Brain Death Organ Donors: a Randomized Controled Trial
Acronym: ECHOT4
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment was too slow and we cannot anticipate to recruit the target sample size
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Responsible Party: Principal Investigator, Anne Julie Frenette, Intensive Care Pharmacist, Associate Clinical Professor, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2014-987
Record Dates: First submitted 2014-08-01; First posted 2014-08-07 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Brain Dead Organ Donors
Keywords: Organ donation; Brain dead; Levothyroxine
MeSH Terms: conditions — Brain Death | interventions — Thyroxine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levothyroxine (Active Comparator): Levothyroxine infusion 20 mg IV bolus then 10 mg/h infusion
  Interventions: Drug: Levothyroxine
- Placebo (Placebo Comparator): Infusion matched to intervention arm
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Levothyroxine — 20 mg IV bolus + 10 mg/h infusion
  Other Names: Synthroid(R)
  Arms: Levothyroxine
Drug: placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the feasibility of a randomized controlled trial comparing levothyroxine to placebo in neurologically deceased donors

ELIGIBILITY:
Inclusion Criteria:

* Prior signed written informed from family member (no more needed following amendment in July 2016)
* 16 years of age or older
* Brain death diagnosis
* Left ventricular ejection fraction < 50% determined by transthoracic echocardiography or hemodynamic instability defined as a mean dose of noradrenaline 0.1 mcg/kg/min + vasopressin

Exclusion Criteria:

* Heart failure history (removed after june 2015)
* Chronic exogenous oral T4 or T3 before death (removed after june 2015)
* Having received T4 infusion before recruitment(removed after june 2015)
* Echographic images not interpretable

  * Age 75 and older(removed after june 2015)
  * Prior coronary heart disease defined as prior coronary artery bypass graft or percutaneous coronary intervention (with or without stents)(removed after june 2015)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Study feasibility | In 2 years
  1) proportion of eligible recruited patients 2)proportion of recruited patients who completed the study 3) proportion of protocol violation
Variation in left ventricular ejection fraction | 6 hours post infusion

SECONDARY OUTCOMES:
Numbers of donated hearts | On organ donation surgery
Incidence of de novo atrial fibrillation | From beginning of infusion until beginning of retrieval surgery
Time from recruitment to the administration of the study drug | From randomization to 12 hours post randomization

CONTACTS AND LOCATIONS:
Overall Officials: Anne Julie Frenette, M.Sc, Principal Investigator — Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Locations (1):
- Hopital du Sacré-Coeur de Montreal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Frenette AJ, Williamson D, Williams V, Lagace AM, Charbonney E, Serri K. A Pilot Randomized Controlled Trial Comparing Levothyroxine to Placebo in Neurologically Deceased Donors. Prog Transplant. 2019 Sep;29(3):261-268. doi: 10.1177/1526924819855083. Epub 2019 Jun 9. PMID 31179831